CLINICAL TRIAL: NCT07141524
Title: Ventilation-Perfusion Matching and PEEP Titration in Patients Undergoing Peripheral Veno-Arterial Extracorporeal Membrane Oxygenation (VA ECMO)
Brief Title: Optimizing Breathing and Blood Flow in Patients Treated With VA ECMO
Acronym: ECMO-VP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Maurizio Bottiroli, Assistant Professor of Anesthesia, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2025P000675
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-10

CONDITIONS: VA-ECMO
Keywords: Ventilation / perfusion; ECMO; Mechanical Ventilation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lung physiology assessment (Other): Measurement of lung perfusion (via EIT) and transpulmonary pressure (via esophageal manometry) during decremental PEEP trial
  Interventions: Other: Physiology measurements

INTERVENTIONS:
Other: Physiology measurements — Measurement of lung perfusion (via EIT) and transpulmonary pressure (via esophageal manometry) during decremental PEEP trial

SUMMARY:
The aim of this study is to characterize ventilation/perfusion (V/Q) matching in adult patients receiving peripheral VA ECMO support while on mechanical ventilation, and to evaluate the impact of PEEP titration guided by Electrical Impedance Tomography (EIT) and esophageal pressure measurements on lung mechanics and V/Q optimization.

DETAILED DESCRIPTION:
The investigators hypothesize that an individualized PEEP titration guided by esophageal pressure measurements and Electrical Impedance Tomography can reduce lung overdistention, enhance lung recruitment, and improve V/Q matching by optimizing regional ventilation and perfusion also in VA ECMO.

Our objectives are:

1. To describe V/Q matching in patients undergoing mechanical ventilation during peripheral VA ECMO support.
2. To explore the impact of PEEP titration based on esophageal pressure and EIT in terms of lung mechanics and V/Q matching.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) undergoing mechanical ventilation during peripheral VA ECMO support for cardiogenic shock, cardiac arrest, or refractory heart failure.
* On ECMO support for at least 6 hours
* Swan-Ganz catheter required as standard clinical care
* Clinically stable in the estimation of the study investigator

Exclusion Criteria:

* Contraindications to EIT (e.g., presence of pacemaker or IMPELLA device for electrical interference)
* Patients without pulmonary flow (non-pulsatile pulmonary prSessure)
* Patients with known pulmonary embolism
* Imminent withdrawal of life support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
V/Q match | 1 hour
  Primary outcome measure:
  Reduction in shunt fraction (expressed in %)
  Secondary outcome measure:
  Reduction in dead space (expressed as volume)
  Respiratory mechanics will be recorded before and after best PEEP. Ventilation (L/min)/Perfusion (L/min) [V/Q] ratio comparing baseline with best PEEP (after PEEP optimization trial).

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided